CLINICAL TRIAL: NCT02390024
Title: Influence of Persistent Patient / Ventilator Decoupling in Cognitive and Psychopathological Sequelae in Critically Ill Patients: A Multicenter Clinical and Mechanisticstudy
Brief Title: Influence of Patient/Ventilador Decoupling in Neurocognitive and Psychopathological Sequelae in ICU Patients
Acronym: PVI-NCOG
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Althaia Xarxa Assistencial Universitària de Manresa (Other); Hospital Mutua de Terrassa (Other)
Responsible Party: Principal Investigator, Lluis Blanch, Director of the Fundació Parc Taulí, Corporacion Parc Tauli
Other Study IDs: PI13/02204
Record Dates: First submitted 2015-02-27; First posted 2015-03-17 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Critical Illness
Keywords: Mechanical Ventilation; Asynchronies; Cognition
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Critically ill patients: Mechanical Ventilation
  Interventions: Device: Invasive Mechanical Ventilation

INTERVENTIONS:
Device: Invasive Mechanical Ventilation — Mechanical ventilation parameters will be monitorized during the ICU stay in all patients Four types of ventilators will be used:
  Servo Dräger Evita XL Dräger Evita 4 Puritan Bennet 840
  Other Names: Asynchronies

SUMMARY:
Mechanical ventilation (MV) is a vital support tool for critically ill patients. However, it may present several adverse effects, such as the development of cognitive and psychopathological alterations. Patient-ventilator asynchronies occur frequently since the beginning of the MV. These asynchronies are associated with poor clinical outcome and could be responsible for the neuronal changes causing these alterations. The objective of this project is to analyze the influence of patient-ventilation asynchronies in the development of long-term cognitive/psychopathological impairments and to explore the molecular mechanisms that could explain of these alterations. An exploratory, observational, multicenter, non-interventionist study will be performed in 150 ICU patients. The continuous recording of asynchronies and other clinical variables during ICU stay and the results of neuropsychological assessments will enable to identify clinical clusters associated with cognitive/psychopathological impairments.

DETAILED DESCRIPTION:
MV parameters, as well as other physiological variables, will be monitorized during the ICU stay in all patients. A neurocognitive and psychopathological assessment will be administed in all patients at 1-month and 1-year follow up.

After data collection, an asynchronies index will be calculated. A clusters analysis, based on clinical variables and asynchronies index, will be performed. The relationship between patients' clusters and the neuropsychological/ psychopathological data will be analized.

CLINICAL STUDY Univariate descriptive analysis: for quantitative variables the mean, standard deviation, percentiles 25, 50 and 75, minimum is calculated and maximum. For qualitative variables, the absolute and relative frequencies were calculated. Population interval will be estimated at 95% confidence level.

Multivariate analysis: cluster analysis, with the intention to investigate possible associations of individuals and characterization of the profile of each cluster. Comparison of standardized scores (z) of the neuropsychological variables and asynchronies index between clusters will be carried out by parametric or nonparametric techniques, as more appropriate.

Association of asynchrony with the neuropsychological variables: conditional logistic regression (case-control) of the scores of neuropsychological variables (dichotomized) versus asynchronies index will be performed, controlling for confounding covariates or factors that may have a modifier effect. The multivariate case-control matching will be performed by the method of propensity score or by genetic algorithms. The odds ratio and confidence interval of 95% was estimated.

Sample size: has been used rule of thumb for logistic regression models include between 10-15 cases per covariate. In this case, the sample will consist of 150 patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years old.
* No neurological disease
* No evidence of COPD.
* Patients within the following 24 hours at endotracheal intubation and who are clinically expected to receive > 72 hours of mechanical ventilation

Exclusion Criteria:

* No authorization of the family or patient inclusion.
* Age outside the limits.
* Patients with prior neurological disease or focal brain damage prior to admission to the ICU
* Patients with serious psychiatric illness or mental retardation.
* Time monitoring of asynchrony < 80% of the total duration of mechanical ventilation.
* Patients who develop secondary complications (infections, stroke, brain damage or structural TC acquired) after discharge from ICU (during hospital stay) that could compromise the results of neuropsychological assessment.
* Patients with moderate to severe cognitive impairment previous to ICU stay (Short form IQCODE > 57 score)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients undergoing mechanical ventilation and monitored with and advanced continuous monitoring system.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2015-06; Primary Completion 2018-03 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Short-term neurocognitive alterations | 1month after ICU discharge
  This outcome will be a composite outcome measured by:
  Attention / Verbal Working Memory: Digits subtest WAIS III Attention / Visual Working Memory: Spatial Span subtest of the WMS III Verbal Learning and Memory: Auditory Verbal Learning Test Speed of Information Processing: Symbol Search subtest of WAIS III Sequencing and alternating stimuli: Trail Making Test Inhibition of the automatic reply: Stroop Test Verbal Fluency: FAS Semantic Verbal Fluency: Animals 1'

SECONDARY OUTCOMES:
Long-term neurocognitive alterations | 1year after ICU discharge
  This outcome will be a composite outcome measured by::
  Attention / Verbal Working Memory: Digits subtest WAIS III Attention / Visual Working Memory: Spatial Span subtest of the WMS III Verbal Learning and Memory: Auditory Verbal Learning Test Speed of Information Processing: Symbol Search subtest of WAIS III Sequencing and alternating stimuli: Trail Making Test Inhibition of the automatic reply: Stroop Test Verbal Fluency: FAS Semantic Verbal Fluency: Animals 1'
Short-term anxiety and depression symptoms | 1month after ICU discharge
  Measured by::
  Hospital Anxiety and Depression Scale (HADS)
Short-term Post-traumatic Stress Disorder | 1month after ICU discharge
  Measured by:
  Post Traumatic Stress Syndrome: Davidson Trauma Scale
Long-term anxiety and depression symptoms | 1year after ICU discharge
  Measured by:
  Hospital Anxiety and Depression Scale (HADS)
Long-term Post-traumatic Stress Disorder | 1year after ICU discharge
  Measured by:
  Post Traumatic Stress Syndrome: Davidson Trauma Scale

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Blanch Torra, PhD, Principal Investigator — Fundació Parc Taulí
Locations (1):
- Corporación Sanitaria Parc Taulí, Sabadell, Barcelon, Spain

REFERENCES:
- [Derived] Fernandez-Gonzalo S, Navarra-Ventura G, Bacardit N, Goma Fernandez G, de Haro C, Subira C, Lopez-Aguilar J, Magrans R, Sarlabous L, Aquino Esperanza J, Jodar M, Rue M, Ochagavia A, Palao DJ, Fernandez R, Blanch L. Cognitive phenotypes 1 month after ICU discharge in mechanically ventilated patients: a prospective observational cohort study. Crit Care. 2020 Oct 21;24(1):618. doi: 10.1186/s13054-020-03334-2. PMID 33087171